CLINICAL TRIAL: NCT02859376
Title: Analgesic Efficacy of Different Doses of Sucrose During Blood Sampling in Preterm Infants: Prospective, Randomized, Controlled, Double Blind, Clinical Trial
Brief Title: Analgesic Efficacy of Different Doses of Sucrose During Blood Sampling in Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Teresa Mion, MD, University Hospital Padova
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AOP0066025
Record Dates: First submitted 2015-12-16; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Pain
Keywords: Preterm infants; Pain; Sucrose
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sucrose24% 2 minutes before (Active Comparator): sucrose 24% 0,3 mL if < 1000 g or 0,5 mL if > 1000 g two minutes BEFORE the skin breaking procedure
  Interventions: Dietary Supplement: sucrose 24%
- sucrose24% 2minutes before and during (Experimental): sucrose 24% 0,3 mL if < 1000 g or 0,5 mL if > 1000 g two minutes BEFORE and DURING the skin breaking procedure
  Interventions: Dietary Supplement: sucrose 24%

INTERVENTIONS:
Dietary Supplement: sucrose 24% — Premature neonates undergoing blood samples through skin breaking procedures, meeting inclusion criteria, will be randomized as soon as the doctor decision to drown the blood is made, to either sucrose 24% 0,3 mL if < 1000 g or 0,5 mL if > 1000 g two minutes BEFORE the skin breaking procedure or sucrose 24% 0,3 mL if < 1000 g or 0,5 mL if > 1000 g two minutes BEFORE and DURING the skin breaking procedure, according to a computer generated randomization list.

SUMMARY:
The objective of this trial is to compare the analgesic effect of a single dose of oral sucrose 24% administered two minutes before a blood sampling (either heel prick or vascular puncture) versus multiple doses of oral sucrose 24% administered two minutes before and during the procedure in a population of preterm newborns of Gestational Age ≤ 36+6 weeks hospitalized in Neonatal Intensive Care Unit, using neonatal pain scales (Premature Infant Pain Profile (PIPP), Face, Legs, Activity, Cry, Consolability (FLACC) and indirect Visual Analogue Scale (VAS)) and Skin Conductance (SC) measurement (Pain Monitor).

DETAILED DESCRIPTION:
This is a controlled, randomized, double blind, (double--dummy) study to evaluate the analgesic efficacy of sucrose. The study staff will evaluate all inborn newborns admitted to the Neonatal Intensive Care Unit (NICU) with a Gestational Age (GA) ≤36+6 weeks; the newborns will be immediately screened for eligibility based upon the pre--defined study inclusion/exclusion criteria.

Then, the parents will be informed about the study and the written informed consent form will be signed. Those eligible will be randomized into the study through computer generated randomization list.

The population of the study consists of premature infants undergoing blood sampling. It is estimated that approximately 144 premature neonates (72 per group either heel prick or venepuncture) will be included in the randomized study.

All eligible neonates whose parents have agreed to participate in the study by signing the informed consent form will be randomized as soon as they are admitted to the NICU.

This study will be conducted in 3 phases:

* Pre--randomization The following items will be obtained: Maternal history including the mother's medical and pregnancy history, prenatal care status; Antenatal analgesics and sedative drugs given to the mother; Estimated GA, birth weight and length. All the data have to be noted on the Case Report Form (CRF);
* Study phase: Premature neonates undergoing blood samples through skin breaking procedures, meeting inclusion criteria, will be randomized as soon as the doctor decision to drown the blood is made, to either sucrose 24% 0,3 mL if ≤ 1000 g or 0,5 mL if > 1000 g two minutes before the skin breaking procedure or sucrose 24% 0,3 mL if ≤ 1000 g or 0,5 mL if > 1000 g two minutes before and during the skin breaking procedure, according to a computer generated randomization list. A trained operator (a nurse or a doctor) will perform heel pricks using an automatic lance (Tenderfoot® micro--preemie for infants < 1000 g and Tenderfoot preemie for infants > 1000 grams) and venipuncture using a butterfly needle 23--25 gauge. Any skin breaking procedure, either heel prick or venipuncture, for each patient will be noted down;; patients will be video--recorded during blood sampling to allow at least two operators to evaluate the analgesic efficacy of the intervention by algometric measurements. In a subgroup of patients skin conductance will also be measured.

Algometric measurements: The pain evaluation will be done visualizing the video of the procedure. Two different evaluators independently will assign the pain score with:

1. Premature Infant Pain Profile (PIPP) at 30 and 60 seconds after the skin puncture
2. Face, Legs, Activity, Cry, Consolability (FLACC) scale at 30 seconds
3. Indirect Visual Analogue Scale (VAS) at 30 seconds for inter--rater agreement. One week later the same evaluators will assign again the pain scores for the intra--rater agreement.

Instrumental PAIN examinations: Pain Monitor is an instrument that measures SC. It detects hand or foot skin conductance gradient, which is directly related to the painful stimuli. The sympathetic nervous system releases acetylcholine that acts on muscarine receptors inducing a sweating and SC increase in response to painful stimuli. Pain monitor is simple to use: tree electrodes positioned on neonate foot sole are connected to the central system. Pain monitor immediately and continuously reacts to stimuli without being influenced neither by hemodynamic variability nor by neuromuscular blocks. The measurement its represented on a compatible computer monitor through a graphic function with SC values expressed in microsiemens on the ordinate axis and time on the abscissa axis. Stressful and painful stimuli related SC variability is represented by peaks and the under peaks area defines pain intensity at detection moment. During monitoring you can note down directly on the graphic every intervention on the patient (medication, blood sample, ect.). Detection can be extrapolated with Excel for statistical analysis.

- Follow--up phase: it will begin from the end of the blood samples. Assessments will continue until hospital discharge.

AE that are ongoing during the study phase as well as clinical outcomes (that are major clinical diagnoses) will be assessed until hospital discharge. Clinical data will be recorded on CRF. In addition the following information will be collected at hospital discharge:

* Number of previous skin breaking procedures
* Number of previous sucrose doses
* Clinical status of the infant
* Duration of hospitalization
* Number of Ventilated Days
* Need for oxygen/monitor at discharge
* Need for supplemental oxygen at 36 weeks post--menstrual age

ELIGIBILITY:
Inclusion Criteria:

* preterm neonates with gestational age ranging from 23+ 0 to 36+ 6 weeks
* undergoing blood sampling (either heel prick or vascular puncture)
* age ≤ 40 week GA + 28 days at the time of blood sampling
* parental written informed consent for participation in the study must be obtained

Exclusion Criteria:

* Evidence of severe birth asphyxia, that is an APGAR score below 5 at 5 minutes of age and/or umbilical arterial pH < 7.0
* Known genetic or chromosomal disorders
* Myopathies and neuropathies interfering with pain assessment by pain scales
* Sedation
* Presence of central catheter allowing blood sampling without skin breaking
* Other painful procedure less than 2 hours before blood sampling
* Physiological instability (more than 6 episodes of bradycardia and/or apnea per day)
* Maternal drug abuse

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change of analgesic efficacy Premature Infant Pain Profile (PIPP) | 2 minutes before, at the moment of the skin puncture, and at 30, 60 and 120 seconds after the skin puncture
  The primary outcome of this study will be to evaluate the analgesic efficacy of sucrose 24% administration (single versus multiple doses) during blood sampling using Premature Infant Pain Profile (PIPP).

SECONDARY OUTCOMES:
Change of analgesic efficacy Face, Legs, Activity, Cry, Consolability (FLACC) | at 30 and 120 seconds after the skin puncture
  The analgesic efficacy of sucrose 24% administration (single Vs multiple doses) during blood sampling using Face, Legs, Activity, Cry, Consolability (FLACC)
Change of analgesic efficacy Visual Analogue Scale (VAS) | at 30 and 120 seconds after the skin puncture
  The analgesic efficacy of sucrose 24% administration (single Vs multiple doses) during blood sampling using indirect Visual Analogue Scale (VAS).
Change of analgesic efficacy Pain Monitor (skin electrical conductance) | 2 minutes before, at the moment of the skin puncture, and at 30, 60 and 120 seconds after the skin puncture
  The analgesic efficacy of sucrose 24% administration (single Vs multiple doses) during blood sampling using Pain Monitor (skin electrical conductance)
Pain evaluation during heel prick Vs vascular puncture PIPP | Through study completion, an average of 1 year
  Pain evaluation during heel prick Vs vascular puncture will be performed using PIPP scale
Pain evaluation during heel prick Vs vascular puncture FLACC | Through study completion, an average of 1 year
  Pain evaluation during heel prick Vs vascular puncture will be performed using FLACC scale
Pain evaluation during heel prick Vs vascular puncture VAS | Through study completion, an average of 1 year
  Pain evaluation during heel prick Vs vascular puncture will be performed using VAS scale
Pain evaluation during heel prick Vs vascular puncture Pain Monitor (skin electrical conductance) | Through study completion, an average of 1 year
  Pain evaluation during heel prick Vs vascular puncture will be performed using Pain Monitor (skin electrical conductance)
Intra--hospital outcome Mechanical Ventilation (MV) duration | Through study completion, an average of 1 year
  Intra--hospital outcome MV duration
Intra--hospital outcome non-Invasive MV (nIMV) duration | Through study completion, an average of 1 year
  Intra--hospital outcome nIMV duration
Intra--hospital outcome oxygen dependence duration | Through study completion, an average of 1 year
  Intra--hospital outcome oxygen dependence
Intra--hospital outcome rate of Bronchopulmonary Dysplasia (BPD) | Through study completion, an average of 1 year
  Intra--hospital outcome rate of BPD
Intra--hospital outcome rate of Pneumothorax (PNX) | Through study completion, an average of 1 year
  Intra--hospital outcome rate of PNX
Intra--hospital outcome rate of Patent ductus arteriosus (PDA) | Through study completion, an average of 1 year
  Intra--hospital outcome rate of PDA
Intra--hospital outcome incidence Intraventricular hemorrhage (IVH)/ Periventricular leukomalacia (PVL) | Through study completion, an average of 1 year
  Intra--hospital outcome incidence of IVH/PVL
Intra--hospital outcome incidence death within 28 days of life | within 28 days of life
  Intra--hospital outcome incidence of death within 28 days of life
Intra--hospital outcome incidence hydrocephalus | Through study completion, an average of 1 year
  Intra--hospital outcome incidence of hydrocephalus
Intra--hospital outcome time to Full Enteral Feeding (FEF) | Through study completion, an average of 1 year
  Intra--hospital outcome time to FEF
Intra--hospital outcome rate of Necrotizing Enterocolitis (NEC) | Through study completion, an average of 1 year
  Intra--hospital outcome rate of NEC (all stages according to the modified Bell's criteria)
Intra--hospital outcome rate of proved sepsis | Through study completion, an average of 1 year
  Intra--hospital outcome rate of proved sepsis
Intra--hospital outcome rate of suspected sepsis | Through study completion, an average of 1 year
  Intra--hospital outcome rate of suspected sepsis
Intra--hospital outcome rate of Retinopathy of Prematurity (ROP) | Through study completion, an average of 1 year
  Intra--hospital outcome rate of ROP
Intra--hospital outcome time to regain birth weight | Through study completion, an average of 1 year
  Intra--hospital outcome time to regain birth weight
Intra--hospital outcome hospitalization length | Through study completion, an average of 1 year
  Intra--hospital outcome hospitalization length
Intra--hospital outcome incidence hospital discharge without major morbidities | Through study completion, an average of 1 year
  Intra--hospital outcome incidence of hospital discharge without major morbidities
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Through study completion till patient discharge, an average of 1 year
  Safety [achieved by monitoring and registering adverse events (AEs), serious adverse events (SAEs) even those unexpected (SUSARs), and measuring vital signs]

CONTACTS AND LOCATIONS:
Overall Officials: Paola Lago, MD, Principal Investigator
Locations (1):
- University Hospital of Padova, Padua, Padova, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cignacco EL, Sellam G, Stoffel L, Gerull R, Nelle M, Anand KJ, Engberg S. Oral sucrose and "facilitated tucking" for repeated pain relief in preterms: a randomized controlled trial. Pediatrics. 2012 Feb;129(2):299-308. doi: 10.1542/peds.2011-1879. Epub 2012 Jan 9. PMID 22232305
- [Background] Shah PS, Herbozo C, Aliwalas LL, Shah VS. Breastfeeding or breast milk for procedural pain in neonates. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD004950. doi: 10.1002/14651858.CD004950.pub3. PMID 23235618
- [Background] Simonse E, Mulder PG, van Beek RH. Analgesic effect of breast milk versus sucrose for analgesia during heel lance in late preterm infants. Pediatrics. 2012 Apr;129(4):657-63. doi: 10.1542/peds.2011-2173. Epub 2012 Mar 5. PMID 22392168
- [Background] Yin T, Yang L, Lee TY, Li CC, Hua YM, Liaw JJ. Development of atraumatic heel-stick procedures by combined treatment with non-nutritive sucking, oral sucrose, and facilitated tucking: a randomised, controlled trial. Int J Nurs Stud. 2015 Aug;52(8):1288-99. doi: 10.1016/j.ijnurstu.2015.04.012. Epub 2015 Apr 23. PMID 25939641
- [Background] Shah VS, Ohlsson A. Venepuncture versus heel lance for blood sampling in term neonates. Cochrane Database Syst Rev. 2011 Oct 5;2011(10):CD001452. doi: 10.1002/14651858.CD001452.pub4. PMID 21975734
- [Background] Stevens B, Yamada J, Lee GY, Ohlsson A. Sucrose for analgesia in newborn infants undergoing painful procedures. Cochrane Database Syst Rev. 2013 Jan 31;(1):CD001069. doi: 10.1002/14651858.CD001069.pub4. PMID 23440783